CLINICAL TRIAL: NCT02058706
Title: Randomized Phase II Screening Trial of Enzalutamide/MDV-3100 and LHRH Analogue vs Combined Androgen Deprivation (LHRH Analogue + Bicalutamide) in Metastatic Hormone Sensitive Prostate Cancer
Brief Title: LHRH Analogue Therapy With Enzalutamide or Bicalutamide in Treating Patients With Hormone Sensitive Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elisabeth Heath, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-083; NCI-2014-00212 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-083 (Other: Barbara Ann Karmanos Cancer Institute); P30CA022453 (NIH)
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Results first posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; bicalutamide; Orchiectomy; Leuprolide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (enzalutamide and LHRH analogue therapy) (Experimental): Patients receive enzalutamide orally PO QD and undergo orchiectomy or receive LHRH analogue therapy (leuprolide acetate, goserelin acetate, or any other FDA approved preparation). Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: enzalutamide; Procedure: orchiectomy; Drug: leuprolide acetate; Drug: goserelin acetate; Other: laboratory biomarker analysis
- Arm B (bicalutamide and LHRH analogue therapy) (Active Comparator): Patients receive bicalutamide PO QD and undergo orchiectomy or receive LHRH analogue therapy as in Arm A. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bicalutamide; Procedure: orchiectomy; Drug: leuprolide acetate; Drug: goserelin acetate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: enzalutamide — Given PO
  Other Names: MDV3100; selective androgen receptor modulator MDV3100; XTANDI
  Arms: Arm A (enzalutamide and LHRH analogue therapy)
Drug: bicalutamide — Given PO
  Other Names: Casodex; CDX
  Arms: Arm B (bicalutamide and LHRH analogue therapy)
Procedure: orchiectomy — Undergo orchiectomy or receive LHRH analogue therapy
Drug: leuprolide acetate — Undergo orchiectomy or receive LHRH analogue therapy
  Other Names: Enantone; LEUP; Lupron; Lupron Depot
Drug: goserelin acetate — Undergo orchiectomy or receive LHRH analogue therapy
  Other Names: ICI-118630; ZDX; Zoladex
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies if enzalutamide added to standard luteinizing hormone-releasing hormone (LHRH) analogue therapy will improve effects against prostate cancer compared to the standard therapy of LHRH analogue and bicalutamide. Hormone therapies stop the body from producing or block the effect of male sex hormones (testosterone). Enzalutamide blocks the effect of male sex hormones which are responsible for the growth of prostate cancer. Hormonal therapies that lower the level of testosterone are among the most effective treatments for prostate cancer that have spread to other areas of the body (metastasized). It is not yet known whether LHRH analogue therapy with bicalutamide is more effective than LHRH analogue therapy with enzalutamide in treating prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the rates of achieving prostate-specific antigen (PSA) remission at month 7 with LHRH analogue therapy and enzalutamide (Arm A) with that achieved with LHRH analogue and bicalutamide (Arm B) in metastatic hormone sensitive prostate cancer.

SECONDARY OBJECTIVES:

I. To compare the primary endpoint by race. II. To compare the rates of each of 2 types of response by treatment arm: measurable disease response; and PSA response.

III. To compare each of 7 time-to-event endpoints by treatment arm: duration of overall response (RD); duration of stable disease (SDD); time to treatment failure (TTF); time-to-progression (TTP); TTP in patients with bone metastases; progression-free survival (PFS); and overall survival (OS).

IV. To compare the rates of each type of toxicity by treatment arm. V. To compare the incidence rate of skeletal related events (SRE), and the time until SRE, separately by treatment arm.

VI. To compare the rates of circulating tumor cell (CTC) response by treatment arm.

VIII. To explore the molecular mechanisms within the androgen receptor pathway by determining the levels of chemokine (C-X-C motif) receptor 4 (CXCR4) and transmembrane protease, serine 2 (TMPRSS2)-v-ets avian erythroblastosis virus E26 oncogene homolog (ERG) expression, androgen metabolism enzymes; androgen receptor variants, and length of cytosine-adenine-guanine (CAG) repeats within the androgen receptor gene, and to associate them with the primary endpoint.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive enzalutamide orally (PO) once daily (QD) and undergo orchiectomy or receive LHRH analogue therapy (leuprolide acetate, goserelin acetate, or any other Food and Drug Administration [FDA] approved preparation). Treatment continues in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive bicalutamide PO QD and undergo orchiectomy or receive LHRH analogue therapy as in Arm A. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma with metastasis either starting or recently started on LHRH analogue therapy. [Late induction permitted within 3 months of starting LHRH analogue therapy or antiandrogen]
* All patients who have not initiated hormone therapy (Early induction patients) must have elevated PSA ≥ 4 ng/ml within 28 days prior to registration. For late induction registrations, PSA must be ≥ 4 ng/ml prior to start of androgen deprivation therapy; either antiandrogen or LHRH analogue or GNRH antagonist .If patients are on antiandrogen, this will need to be discontinued for at least 7 days prior to registration.
* Patients with a history of prior neoadjuvant or adjuvant hormone therapy are eligible provided they have received twenty four or less months of hormone treatment (single or combination treatment, excluding orchiectomy). Both therapies (neoadjuvant/adjuvant hormone therapy) must have been discontinued at least 6 months prior to registration. This is intended to exclude patients who might have been rendered indirectly androgen insensitive.
* There must be no plans to receive concomitant chemotherapy, biological response modifiers, radiation therapy or hormonal therapy. Concomitant radiation therapy is allowed for the palliation of severe pain/neuropathic compression. Prior or concomitant use of megestrol acetate for the treatment of hot flashes is allowed.
* Patients must have a performance status of 0 - 2 by Zubrod Criteria.
* Patients must have recovered from any major infections and/or surgical procedures and,in the opinion of the investigator, not have significant active medical illness precluding protocol treatment or survival.
* No prior malignancy is allowed except for adequately treated basal cell (or squamous cell) skin cancer, superficial or in situ cancer of the bladder. For an invasive cancer the patients should be disease free for at least 3 years prior to enrollment on study.
* For all patients a bone scan must be performed within 60 days prior to registration for tumor assessment. CT scans (abdomen and pelvis) and chest x-ray are optional, but must be repeated if used for disease assessment. For late induction registrations, tumor assessment imaging showing metastatic disease must be available prior to start of androgen deprivation therapy.
* Age 18 or older and willing and able to provide informed consent.
* Willingness to swallow pills and no medical condition that would interfere with this.
* Male patient and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (one of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 3 months after final study drug administration. Patients are also required to use a condom if having sex with a pregnant woman.
* Patient should agree to a tumor tissue biopsy prior to protocol enrollment. Post therapy biopsy is optional.
* Patients who are being treated with a GNRH antagonist should be willing to switch to a LHRH analogue after registration.
* Patients must have one of the following a) Low volume disease (defined as no visceral metastases and < 4 bone metastases) or b) are not candidates for docetaxel based chemotherapy or 3) refused docetaxel chemotherapy

Exclusion Criteria:

* History of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke, significant brain trauma) at any time in the past. Also, history of loss of consciousness or transient ischemic attack within 12 months of Day 1 visit;
* Known or suspected brain metastasis or active leptomeningeal disease;
* Severe concurrent disease, infection, or co-morbidity that, in the judgment of the Investigator, would make the patient inappropriate for enrollment;
* Absolute neutrophil count < 1,000/μL, or platelet count < 50,000/μL, or hemoglobin<8 g/dL) at the Screening visit.
* Total bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times the upper limit of normal
* Creatinine > 177 μmol/L (2 mg/dL)
* Clinically significant cardiovascular disease including: Myocardial infarction within 6 months; Uncontrolled angina within 3 months; Congestive heart failure New York Heart Association (NYHA) class 3 or 4, or patients with history of congestive heart failure (NYHA) class 3 or 4 in the past, unless screening echocardiogram or multi-gated acquisition scan performed within 3 months results in a left ventricular ejection fraction that is greater or equal to 45%; History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes); History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place; Hypotension as indicated by systolic blood pressure < 86 millimeters of mercury (mmHg) at the Screening visit; Bradycardia as indicated by a heart rate of < 50 beats per minute on the Screening ECG; Uncontrolled hypertension as indicated by systolic blood pressure > 170 mmHg or diastolic blood pressure > 105 mmHg
* Gastrointestinal disorder affecting absorption (e.g., gastrectomy, active peptic ulcer disease within last 3 months);
* Treatment with concurrent 5-α reductase inhibitors (finasteride, dutasteride), estrogens, and/or cyproterone
* Treatment with systemic biologic therapy for prostate cancer (other than approved bone targeted agents and GnRH-analogue therapy) or other agents with anti-tumor activity within 4 weeks of enrollment (Day 1 visit);
* History of prostate cancer progression on ketoconazole;
* Prior use, or participation in a clinical trial, of an investigational agent that blocks androgen synthesis (e.g., abiraterone acetate, TAK-700, TAK-683, TAK-448) or agents that block the androgen receptor (e.g.,ARN-509)
* Previous enzalutamide therapy;
* Use of an investigational agent within 2 weeks of enrollment (Day 1 visit);
* Use of herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease PSA levels (e.g., saw palmetto) or systemic corticosteroids greater than the equivalent of replacement steroids or > equivalent of 10 mg of prednisone per day within 4 weeks of enrollment (Day 1 visit);
* Any condition or reason that, in the opinion of the Investigator, interferes with the ability of the patient to participate in the trial, which places the patient at undue risk, or complicates the interpretation of safety data.
* Prior chemotherapy for metastatic disease.
* >30 days of antiandrogen therapy monotherapy without androgen deprivation therapy.
* Life expectancy of 6 months or less.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-05; Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Heath, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ohio State University Medical Center, Columbus, Ohio

REFERENCES:
- [Derived] Vaishampayan UN, Heilbrun LK, Monk P 3rd, Tejwani S, Sonpavde G, Hwang C, Smith D, Jasti P, Dobson K, Dickow B, Heath EI, Semaan L, Cher ML, Fontana JA, Chinni S. Clinical Efficacy of Enzalutamide vs Bicalutamide Combined With Androgen Deprivation Therapy in Men With Metastatic Hormone-Sensitive Prostate Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jan 4;4(1):e2034633. doi: 10.1001/jamanetworkopen.2020.34633. PMID 33496795

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm B (Bicalutamide and LHRH Analogue Therapy) | Arm A (Enzalutamide and LHRH Analogue Therapy)
Started | 35 | 36
Completed | 35 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Enzalutamide and LHRH Analogue Therapy) | Arm B (Bicalutamide and LHRH Analogue Therapy) | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 18 | 32
  >=65 years | 22 | 17 | 39
Age, Continuous [Median (Full Range); unit: years] | 66 [54 to 86] | 63 [46 to 84] | 65 [46 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 36 | 35 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 14 | 29
  White | 21 | 21 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 35 | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With PSA Remission Assessed Using the Prostate Cancer Clinical Trials Working Group (PCWG2) Criteria
Description: Number of Participants with PSA Remission Assessed Using the Prostate Cancer Clinical Trials Working Group (PCWG2) Criteria specifically at the 7 month time point. The binary endpoint (yes/no) will be summarized with its point estimate (an occurrence rate), and 2-sided Wilson type 95% confidence interval (CI). PSA response rates will be compared by treatment arm in a stratified logistic regression model.
Time Frame: Month 7
Population: Those patients who reached month 7 and had a blood sample tested for PSA at month 7.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Enzalutamide and LHRH Analogue Therapy) | Arm B (Bicalutamide and LHRH Analogue Therapy)
Number analyzed (Participants) | 31 | 24
Participants | 29 | 16

2. Secondary Outcome: Achievement of Measurable Disease Response
Description: The number of participants with Measurable disease response per RECIST v1.1.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Enzalutamide and LHRH Analogue Therapy) | Arm B (Bicalutamide and LHRH Analogue Therapy)
Number analyzed (Participants) | 36 | 35
Participants | 17 | 17

3. Secondary Outcome: Achievement of PSA Response Assessed Using PCWG2 Criteria
Description: Will be summarized with point estimates (occurrence rates), and 2-sided Wilson type 95% CIs.
Time Frame: Up to 2 years
Population: Those patients who reached month 7 of treatment and had a blood sample tested for PSA at any time at or past month 7.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Enzalutamide and LHRH Analogue Therapy) | Arm B (Bicalutamide and LHRH Analogue Therapy)
Number analyzed (Participants) | 32 | 26
Participants | 30 | 17

4. Secondary Outcome: The Percentage of Patients Responding
Description: Point estimates will be calculated and CI estimates will be derived from the Wilcoxon method using STATA software.
Time Frame: 6 months
Measure: Number (90% Confidence Interval); unit: percentage of response at 6 months
Arm/Group | Arm A (Enzalutamide and LHRH Analogue Therapy) | Arm B (Bicalutamide and LHRH Analogue Therapy)
Number analyzed (Participants) | 36 | 35
percentage of response at 6 months | 86 [62 to 95] | 79 [48 to 92]

5. Secondary Outcome: Time to Treatment Failure
Description: Time to Treatment Failure from date of first treatment to date off treatment or date patient is taken off study for any reason. TTF will be estimated with standard K-M methodology. Point and CI estimates of the median and various time point-specific rates will be derived from the K-M life table.
Time Frame: Assessed up to 6 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm B (Bicalutamide and LHRH Analogue Therapy) | Arm A (Enzalutamide and LHRH Analogue Therapy)
Number analyzed (Participants) | 35 | 36
months | 8.2 [5.7 to 11.4] | 20.6 [6.9 to 42.3]

6. Secondary Outcome: Percentage of Patients Progression Free at One Year
Description: Percentage of patients progression free at one year using the Kaplan-Meier method.
Time Frame: assessed at 1 year
Measure: Number (95% Confidence Interval); unit: % participants not progressed at 1 year
Arm/Group | Arm A (Enzalutamide and LHRH Analogue Therapy) | Arm B (Bicalutamide and LHRH Analogue Therapy)
Number analyzed (Participants) | 36 | 35
% participants not progressed at 1 year | 84 [57 to 95] | 34 [15 to 58]

7. Secondary Outcome: Percentage of Patients With Bone Metastases Progression Free at Six Months
Description: Percentage of patients with bone metastases Progression free at six months using the Kaplan-Meier method.
Time Frame: assessed at six months
Population: Patients with bone lesions at baseline.
Measure: Number (95% Confidence Interval); unit: percentage not progressed at 6 months
Arm/Group | Arm A (Enzalutamide and LHRH Analogue Therapy) | Arm B (Bicalutamide and LHRH Analogue Therapy)
Number analyzed (Participants) | 31 | 28
percentage not progressed at 6 months | 91 [63 to 98] | 33 [14 to 54]

8. Secondary Outcome: Percentage of Patients Progression-free at 6 Months
Description: Will be estimated with standard K-M methodology. Point and CI estimates of the six-month rate will be derived from the K-M life table.
Time Frame: From registration to PSA progression defined by PCWG II criteria or measurable disease by RECIST 1.1, assessed at 6 months
Measure: Number (95% Confidence Interval); unit: percentage progression-free at 6 months
Arm/Group | Arm A (Enzalutamide and LHRH Analogue Therapy) | Arm B (Bicalutamide and LHRH Analogue Therapy)
Number analyzed (Participants) | 36 | 35
percentage progression-free at 6 months | 92 [66 to 98] | 45 [25 to 64]

9. Secondary Outcome: Overall Survival at 2 Years
Description: Overall Survival will be measured from date of registration to death or last follow up. OS will be estimated with standard K-M methodology. Point and CI estimates of the 2-year rate will derived from the K-M life table.
Time Frame: Assessed at 2 years
Measure: Number (95% Confidence Interval); unit: percentage alive at 2 years
Arm/Group | Arm A (Enzalutamide and LHRH Analogue Therapy) | Arm B (Bicalutamide and LHRH Analogue Therapy)
Number analyzed (Participants) | 36 | 35
percentage alive at 2 years | 82 [63 to 92] | 54 [34 to 70]

10. Secondary Outcome: The Number of Participants With a CTC Response
Description: Will be summarized with point estimates (occurrence rates). A CTC response is defined as any level of CTC < 5 that is maintained or any level of CTC that is reduced from baseline.
Time Frame: Up to month 1
Population: Patients with sufficient blood sample to test for CTC at baseline and post-treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm B (Bicalutamide and LHRH Analogue Therapy) | Arm A (Enzalutamide and LHRH Analogue Therapy)
Number analyzed (Participants) | 25 | 26
Participants | 17 | 22

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed up to 2 years.
Arm/Group | Arm A (Enzalutamide and LHRH Analogue Therapy) | Arm B (Bicalutamide and LHRH Analogue Therapy)
All-Cause Mortality (participants affected / at risk) | 8/36 | 18/35
Serious Adverse Events (participants affected / at risk) | 17/36 | 16/35
Other Adverse Events (participants affected / at risk) | 33/36 | 33/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Enzalutamide and LHRH Analogue Therapy) (N=36) | Arm B (Bicalutamide and LHRH Analogue Therapy) (N=35)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (General disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fall (General disorders) | 1 (1) | 0 (0)
Fatigue (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Hot flashes (Endocrine disorders) | 0 (0) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 5 (6) | 6 (9)
Hypertriglyceridemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
INR increased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Injection site reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Syncope (Vascular disorders) | 3 (3) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 2 (2) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weight gain (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Weight loss (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Enzalutamide and LHRH Analogue Therapy) (N=36) | Arm B (Bicalutamide and LHRH Analogue Therapy) (N=35)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (5)
Anorexia (General disorders) | 7 (9) | 2 (2)
Anxiety (Psychiatric disorders) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 6 (6)
Blurred vision (Eye disorders) | 3 (3) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (2) | 2 (2)
Confusion (Psychiatric disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (8) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Depression (Psychiatric disorders) | 5 (5) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (12) | 1 (1)
Dizziness (Nervous system disorders) | 8 (14) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 1 (1)
Fall (General disorders) | 3 (4) | 1 (1)
Fatigue (General disorders) | 19 (22) | 10 (11)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (2) | 3 (4)
Headache (Nervous system disorders) | 3 (3) | 6 (8)
Hot flashes (Vascular disorders) | 25 (28) | 20 (23)
Hypertension (Vascular disorders) | 7 (9) | 3 (5)
Hypotension (Vascular disorders) | 2 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 4 (4)
Memory impairment (Nervous system disorders) | 6 (6) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 7 (12) | 4 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2)
Nausea (Gastrointestinal disorders) | 6 (6) | 2 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 5 (7) | 1 (1)
Pain (General disorders) | 13 (18) | 6 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 3 (3) | 3 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 7 (10) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 6 (8) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 3 (5)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 4 (5) | 6 (7)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (4) | 0 (0)
Weight gain (General disorders) | 3 (6) | 4 (9)
Weight loss (Investigations) | 5 (7) | 2 (2)
Edema limbs (General disorders) | 2 (3) | 4 (5)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2) | 5 (7)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT02058706/Prot_SAP_000.pdf